CLINICAL TRIAL: NCT06304207
Title: Comparison of Telehealth and Onsite Supervised Maintenance Exercise Program for Adults With Chronic Lung Disease: A Pilot Randomized Controlled Trial
Brief Title: Telehealth and Onsite Maintenance Exercise in Chronic Lung Disease
Acronym: CLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MGH Institute of Health Professions (Other)
Responsible Party: Principal Investigator, Shweta Gore, Associate Professor, MGH Institute of Health Professions
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 300423
Record Dates: First submitted 2023-06-20; First posted 2024-03-12 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Copd; COPD Exacerbation; COPD Bronchitis; Emphysema or COPD; Chronic Lung Disease; Pulmonary Fibrosis; Interstitial Lung Disease; Bronchiectasis; Chronic Asthma; Chronic Asthmatic Bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Pulmonary Fibrosis; Lung Diseases, Interstitial; Bronchiectasis

STUDY DESIGN:
Intervention Model Description: The study design will be a pilot randomized controlled, assessor-blinded trial with three groups: 1) Tele-rehab where patient will be at home but will receive supervised intervention remotely, 2) Onsite outpatient physical therapy, 3) Control group.
Who Masked: Outcomes Assessor
Masking Description: All baseline and follow up outcomes assessment will be conducted by a study team member blinded to the subject group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Control group participants will only be seen during the outcomes assessments at the MGH Institute of Health Professions at times 0, 1, and 2, but will receive no active supervised intervention. Control group participants will go home with discharge instructions to maintain a home exercise routine provided to them at discharge. Bi-weekly check in phone calls from the study team will continue to ensure participant engagement in the study. During the phone calls, participants will be encouraged to keep a log of their weekly activities in a journal.
- Onsite Pulmonary Rehab (Experimental): Supervised pulmonary rehabilitation including exercise training, activity counselling, and education provided onsite.
  Interventions: Combination Product: Onsite Maintenance Exercise Training
- Telehealth Pulmonary Rehab (Experimental): Supervised pulmonary rehabilitation including exercise training, activity counselling, and education provided remotely using Zoom videoconferencing technology.
  Interventions: Combination Product: Telehealth Maintenance Exercise

INTERVENTIONS:
Combination Product: Onsite Maintenance Exercise Training — Participants will receive a 60-minute supervised weekly exercise intervention for 8-weeks.Each 60-minute session will be broken down into a brief 5-minute training on inspiratory muscle training using a Threshold Inspiratory Muscle Trainer (IMT), 5-minute education on self-management of airway clearance and importance of maintaining regular physical activity; a 5-minute warm-up, and 25 minutes of aerobic training. The training intensity will be derived from the distance covered on the six-minute walk test administered at baseline. Training will be performed at 60-85% of VO2 reserve and converted to walking distance and speed using American College of Sports Medicine walking equations for treadmill and overground walking activities or a corresponding rating of perceived exertion (RPE) of 13-16 for non-walking activities. This will be followed by 15-minutes of functional strength training focusing on the lower extremity muscles, and 5 minutes of cool down with stretching exercises.
  Other Names: Onsite Maintenance Pulmonary Rehab
  Arms: Onsite Pulmonary Rehab
Combination Product: Telehealth Maintenance Exercise — Participants in the tele-rehab group will also receive the same intervention as outlined for the onsite group. The mode of aerobic exercise will vary based on availability of equipment in patient homes. The intervention will be delivered remotely via previously researched models using a tablet computer. I-pads will be provided to the participants on a need basis to take home for the duration of the study. Videoconferencing will be via Partners log in enabled Zoom videoconferencing software (San Jose, California, USA) that allows all participants to see and speak to each other. To ensure safety and understanding of equipment operation and the exercise program, the initial training session and establishment of the home exercise program will occur during the initial onsite visit in the clinic at MGH Institute of Health Professions.
  Other Names: Telehealth Maintenance Pulmonary Rehab
  Arms: Telehealth Pulmonary Rehab

SUMMARY:
The goal of this pilot clinical trial is to compare telehealth and onsite supervised maintenance exercise program for adults with Chronic Lung Disease.

The specific aims of the study are:

* To compare 8-week supervised maintenance program delivered onsite and via tele-rehab with no maintenance for patients with Chronic Lung Disease following discharge from traditional exercise or physical therapy or onsite outpatient rehabilitation programs on clinical outcomes (dyspnea, exercise capacity, physical function, physical activity, and quality of life) at 8 weeks and 4-months post-intervention.
* To compare the differences in dyspnea, exercise capacity, physical function, physical activity, and quality of life between an 8-week maintenance program delivered onsite and via tele-rehab at 8-weeks and 4-months post-intervention in patients with Chronic Lung Disease following discharge from traditional onsite outpatient rehabilitation.

Participants in both intervention groups (onsite and tele-rehab) will undergo a baseline onsite assessment followed by an 8-week supervised exercise intervention either onsite or in a telehealth setting. Control group will receive biweekly check in calls, but no active intervention.

DETAILED DESCRIPTION:
Random Assignment Participants will be randomly assigned using a web-based randomization service (www.randomize.net) to one of three groups: 1) tele-rehab where patient will be at home but will receive supervised intervention remotely, 2) onsite outpatient rehabilitation, and 3) control group, using a computerized random number generator to eliminate risk of bias during allocation.

Subject Enrollment Consent: Potential participants who express interest in the study will be contacted via a phone call by the study team to go over screening and to seek consent for the study. Pre-screening questions will be asked over the phone to confirm eligibility. The letter of informed consent will be read out during the initial phone call and participants will be asked to sign a copy of the consent form prior to their initial visit at the IMPACT Practice Center at MGH Institute of Health Professions via a RedCap link sent to their email. Any questions related to the study will be answered prior to getting a signature on the consent form (See attached consent form). Participants will be informed of the possibility of being in one of three groups. The study Investigators will be involved in obtaining consent. Control group participants will be offered an opportunity to complete an 8-week onsite or tele-rehab intervention upon completion of the study duration. Participants will be able to withdraw from the study at any point with no penalties or any negative consequences. Participation will be voluntary, and participants can choose to step out of the study at any time.

To enhance enrollment of participants from diverse and under-represented backgrounds, free parking will be provided to the onsite location at MGH Institute of Health Professions. For participants assigned to the tele-rehab group, who do not have the means to connect and participate in the intervention, will be loaned an I-pad for the duration of the study. In addition, all participants will be provided with a $50.00 gift card at the end of the study period for their participation in the study.

6. STUDY PROCEDURES

Following informed consent, all participants will undergo a baseline assessment at index date or time point 0. Since the recruitment will occur on a rolling basis, the time 0 will vary for participants.

Outcome Assessments (time 0-time 2)

All outcomes will be recorded at baseline prior to beginning of intervention (time 0), at the end of the study intervention at 8 weeks (time 1), and at 4 months follow-up (time 2) post intervention. Each participant (n=30) will start at time 0 with examination of outcome measurements at the IMPACT practice center at MGH IHP. Outcomes will be assessed by a study team member who will be blinded to the group allocation. Outcomes assessed will include the modified Medical Research Council (mMRC) scale and the dyspnea rating scale for dyspnea, physical function measured by the 30 seconds chair rise test and the 10-meter walk test, functional capacity measured by the six minute walk test, physical activity measured by the International Physical Activity Questionnaire, and quality of life measured by the COPD Assessment Test (CAT) and the PROMIS Global Health Scale Assessment of inspiratory muscle strength will be performed using the maximal inspiratory pressure gauge (MIP). In addition, baseline vitals (heart rate, respiratory rate, oxygen saturation (SpO2) via pulse oximeter, and rating of perceived exertion (RPE) scale at rest will be documented.

The training intensity will be derived from the distance covered on the six-minute walk test. Although participants completing the traditional onsite rehabilitation program at MGH are extensively educated and independent in self-monitoring their oxygen saturation through pulse oximetry, RPE and heart rate, these will be reviewed thoroughly during the initial visit with all participants. In addition to these outcomes, participants will be asked to report any planned or unplanned physician visits, emergency room visits, falls, and injuries. The number of sessions attended by participants will also be recorded.

All participants will receive printed educational resources from the COPD Foundation and Pulmonary Fibrosis Foundation on 1) tips for living well with Chronic Lung Disease, 2) Impact of smoking, and 3) Chronic Lung Disease action plan including resources for disaster preparedness.

Following assessment of outcomes at baseline, participants will begin the 8-week intervention. Supervised visits will occur once every week for both the onsite and tele-rehab groups.

Interventions:

Participants in both intervention groups (onsite and tele-rehab) will receive a 60-minute supervised weekly exercise intervention. Interventions will be delivered by study team members that are licensed physical therapists or students under the supervision of these physical therapists. The study personnel will be paid to provide the intervention and/ collect outcomes. All participants will receive similar interventions as described in Table 1. The interventions received will be similar to standard clinical sessions, however participants and/or their insurers will not be charged for either the on-site or the telehealth interventions.

Each 60-minute session will be broken down into separate sections. These include a brief 5-minute training on inspiratory muscle training using a Threshold Inspiratory Muscle Trainer (IMT), Respironics Threshold PEP and 5-minute check-in a review of their activities during the week at home and any changes in symptoms as well as education on self-management of airway clearance and importance of maintaining regular physical activity. This will be followed by a 5-minute warm-up and 25 minutes of aerobic training in the form of walking, cycling, stair climbing, or NuStep (based on availability and patient preference). The training intensity will be derived from the distance covered on the six-minute walk test administered at baseline. Peak oxygen consumption (VO2) will be estimated based on previously published regression equations. Training will be performed at 60-85% of VO2 reserve and converted to walking distance and speed using American College of Sports Medicine walking equations for treadmill and overground walking activities or a corresponding rating of perceived exertion (RPE) of 13-16 for non-walking activities (cycling, stair climbing). Aerobic training may be completed in shorter intervals if continuous training is limited by symptoms (e.g., 2 × 12.5 minutes or 3 × 8.3 minutes). This will be followed by 15-minutes of functional strength training focusing on the lower extremity muscles such as partial squats, sit to stand exercise, lunges, and step ups and downs.

Progression of exercise will occur each week as: increase in walking or stair climbing speed, increase in wattage of cycle ergometer and NuStep by 5-10% while maintaining dyspnea levels of 3-4/10 on the dyspnea rating scale and maintaining an RPE of 13-16. Functional strengthening exercises will be progressed by increasing number repetitions while maintaining the dyspnea rating scale at 3-4/10. Inspiratory muscle training will progress by 5% each week to maintain dyspnea levels of 3-4/10 on the dyspnea rating scale. If the progression in any of the components elicits dyspnea more than 4, the same training intensity will be continued for another week.

All participants will be encouraged to maintain a log of activities performed during the week.

Tele-rehab group:

Participants in the tele-rehab group will also receive the same intervention as outlined for the onsite group. The mode of aerobic exercise will vary based on availability (see table 1). The intervention will be delivered remotely via previously researched models using a tablet computer. I-pads will be provided to the participants on a need basis to take home for the duration of the study. Videoconferencing will be via Partners log in enabled Zoom videoconferencing software (San Jose, California, USA) that allows all participants to see and speak to each other. To ensure safety and understanding of equipment operation and the exercise program, the initial training session and establishment of the home exercise program will occur during the initial onsite visit in the clinic at MGH Institute of Health Professions.

Although participants completing the traditional onsite rehabilitation program are familiar with and educated on independent in self-monitoring their SpO2, RPE, and heart rate, these will be reviewed during the initial visit with all participants. Pulse oximeters will be provided to participants for the duration of the study.

Fidelity of the exercise training intervention for both groups will be facilitated through regular staff training, and audit of exercise prescription and progression, and assessment of participant engagement.

Control group Control group participants will only be seen during the outcomes assessments at the MGH Institute of Health Professions at times 0, 1, and 2, but will receive no active supervised intervention. Control group participants will go home with discharge instructions to maintain a home exercise routine provided to them at discharge. Bi-weekly check in phone calls from the study team will continue to ensure participant engagement in the study. During the phone calls, participants will be encouraged to keep a log of their weekly activities in a journal.

Data Collection The data that is collected from each patient will include participant demographics (age, sex, comorbidities, body mass index, race, education, work status, living situation (living alone or with partner/caregiver, in independent home or institutionalized), details of interventions provided each visit, log of activities performed during the week, outcome measures, and the number of sessions attended, along with any planned or unplanned physician visits, emergency room visits, hospitalizations, falls, and injuries.

Termination Criteria If a participant is to experience an adverse event during the course of the study, they will be terminated from the study until they receive medical clearance. Adverse events include any falls (with or without injury), hospitalizations, or unplanned visits to their physician for Chronic Lung Disease related symptoms. If patient is unable to return to the study, any data collected up until time of adverse event will be included in study, and the adverse event will be noted. Any adverse events will be reported to the IRB. If patient is allowed to return to regular exercise, the event will still be noted and reported. Any changes in medication or medical status will be monitored.

Remuneration All participants will be given $50.00 in total at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients 40 years and older with physician diagnosed Chronic Lung Disease within 2 months of discharge following completion of a traditional onsite outpatient rehabilitation or physical therapy or exercise program for their condition
* Able to walk independently with or without mobility devices
* Able to complete a six-minute walk test at discharge with or without supplemental oxygen maintaining an oxygen saturation at or above 85%
* Able to follow commands and instructions in the English language
* Have ability to connect to the internet

Exclusion Criteria:

* • Those with significant mobility limitations such as those with a history of stroke, neurological comorbidities such as Parkinson's disease or relapsing multiple sclerosis, or significant degenerative osteoarthritis, or any other joint impairments that compromise ability to walk independently with or without an assistive device.

  * Patients who primarily rely on a wheelchair for mobility
  * Patients with or without supplemental oxygen who are unable to complete a walking test without a drop in oxygen saturation to below 85% at discharge from traditional outpatient rehabilitation
  * Patients with baseline hemodynamic compromise, unstable angina, a recent myocardial infarction within a week, uncontrollable atrial fibrillation not managed with medications, advanced stage heart failure (New York Heart Association class 4), or those with mechanical circulatory assist devices for the heart such a ventricular assist device (VADs)
  * Inability to communicate in the English language

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Exercise Capacity | At baseline
  Exercise capacity as measured by the six-minute walk distance
Exercise Capacity | At 8 weeks (end of the study)
  Exercise capacity as measured by the six-minute walk distance
Exercise Capacity | At 4 months follow up
  Exercise capacity as measured by the six-minute walk distance
Dyspnea | At baseline
  Dyspnea measured on the modified Medical Research Council (mMRC) scale score ranges from 0-4 with higher scores indicating greater shortness of breath
Dyspnea | At 8 weeks (end of the study)
  Dyspnea measured on the modified Medical Research Council (mMRC) scale score ranges from 0-4 with higher scores indicating greater shortness of breath
Dyspnea | At 4 months follow up
  Dyspnea measured on the modified Medical Research Council (mMRC) scale score ranges from 0-4 with higher scores indicating greater shortness of breath
Physical Function | At baseline,
  Physical function measured by the 30 seconds chair rise test
Physical Function | At 8 weeks (end of the study),
  Physical function measured by the 30 seconds chair rise test
Physical Function | At 4 months follow up
  Physical function measured by the 30 seconds chair rise test
Quality of life measure | At baseline
  Quality of life measured by the chronic obstructive pulmonary disease Assessment Test (CAT) scale. Score ranges from 0-40, with higher scores indicating a more severe impact on a patient's life
Quality of life measure | At 8 weeks (end of study)
  Quality of life measured by the chronic obstructive pulmonary disease Assessment Test (CAT) scale. Score ranges from 0-40, with higher scores indicating a more severe impact on a patient's life
Quality of life measure | At 4- month follow up
  Quality of life measured by the chronic obstructive pulmonary disease Assessment Test (CAT) scale. Score ranges from 0-40, with higher scores indicating a more severe impact on a patient's life

SECONDARY OUTCOMES:
Inspiratory muscle strength | At baseline, 8 weeks (end of the study), and at 4 months follow up
  Inspiratory muscle strength assessed via the maximal inspiratory pressure (MIP)
Inspiratory muscle strength | At baseline
  Inspiratory muscle strength assessed via the maximal inspiratory pressure (MIP)
Inspiratory muscle strength | At 8 weeks (end of the study)
  Inspiratory muscle strength assessed via the maximal inspiratory pressure (MIP)
Physical activity | At baseline
  Physical activity measured by the International Physical Activity Questionnaire (IPAQ)
Physical activity | At 8 weeks (end of study)
  Physical activity measured by the International Physical Activity Questionnaire (IPAQ)
Physical activity | At 4 months follow up
  Physical activity measured by the International Physical Activity Questionnaire (IPAQ)
Participants adherence to the program | 8 weeks
  number of sessions attended
Healthcare utilization | 8 weeks
  Number of emergency department visits or unplanned physician visits
Adverse events | 8 weeks
  Falls and/ exacerbations
Patient-Reported Outcomes Measurement Information System (PROMIS) Global 10 score | At baseline
  Quality of life score. It is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient
Patient-Reported Outcomes Measurement Information System (PROMIS) Global 10 score | At 8 weeks (end of study)
  Quality of life score. It is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient
Patient-Reported Outcomes Measurement Information System (PROMIS) Global 10 score | At 4-month follow up
  Quality of life score. It is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient

CONTACTS AND LOCATIONS:
Overall Officials: Shweta Gore, PhD, Principal Investigator — MGH Institute of Health Professions
Locations (1):
- MGH Institute of Health Professions, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
All identifiers will be destroyed and only aggregate data will be shared

REFERENCES:
- [Background] Halbert RJ, Natoli JL, Gano A, Badamgarav E, Buist AS, Mannino DM. Global burden of COPD: systematic review and meta-analysis. Eur Respir J. 2006 Sep;28(3):523-32. doi: 10.1183/09031936.06.00124605. Epub 2006 Apr 12. PMID 16611654
- [Background] 2. American Association of Cardiovascular and Pulmonary Rehabilitation. Guidelines for cardiac rehabilitation and secondary prevention programs. . Champaign, IL: Human Kinetics; 2011.
- [Background] Cruz J, Brooks D, Marques A. Home telemonitoring in COPD: a systematic review of methodologies and patients' adherence. Int J Med Inform. 2014 Apr;83(4):249-63. doi: 10.1016/j.ijmedinf.2014.01.008. Epub 2014 Jan 23. PMID 24529402
- [Background] Rochester CL, Vogiatzis I, Holland AE, Lareau SC, Marciniuk DD, Puhan MA, Spruit MA, Masefield S, Casaburi R, Clini EM, Crouch R, Garcia-Aymerich J, Garvey C, Goldstein RS, Hill K, Morgan M, Nici L, Pitta F, Ries AL, Singh SJ, Troosters T, Wijkstra PJ, Yawn BP, ZuWallack RL; ATS/ERS Task Force on Policy in Pulmonary Rehabilitation. An Official American Thoracic Society/European Respiratory Society Policy Statement: Enhancing Implementation, Use, and Delivery of Pulmonary Rehabilitation. Am J Respir Crit Care Med. 2015 Dec 1;192(11):1373-86. doi: 10.1164/rccm.201510-1966ST. PMID 26623686
- [Background] Bolton CE, Bevan-Smith EF, Blakey JD, Crowe P, Elkin SL, Garrod R, Greening NJ, Heslop K, Hull JH, Man WD, Morgan MD, Proud D, Roberts CM, Sewell L, Singh SJ, Walker PP, Walmsley S; British Thoracic Society Pulmonary Rehabilitation Guideline Development Group; British Thoracic Society Standards of Care Committee. British Thoracic Society guideline on pulmonary rehabilitation in adults. Thorax. 2013 Sep;68 Suppl 2:ii1-30. doi: 10.1136/thoraxjnl-2013-203808. No abstract available. PMID 23880483
- [Background] Marciniuk DD, Brooks D, Butcher S, Debigare R, Dechman G, Ford G, Pepin V, Reid D, Sheel AW, Stickland MK, Todd DC, Walker SL, Aaron SD, Balter M, Bourbeau J, Hernandez P, Maltais F, O'Donnell DE, Bleakney D, Carlin B, Goldstein R, Muthuri SK; Canadian Thoracic Society COPD Committee Expert Working Group. Optimizing pulmonary rehabilitation in chronic obstructive pulmonary disease--practical issues: a Canadian Thoracic Society Clinical Practice Guideline. Can Respir J. 2010 Jul-Aug;17(4):159-68. doi: 10.1155/2010/425975. PMID 20808973
- [Background] Marciniuk DD, Goodridge D, Hernandez P, Rocker G, Balter M, Bailey P, Ford G, Bourbeau J, O'Donnell DE, Maltais F, Mularski RA, Cave AJ, Mayers I, Kennedy V, Oliver TK, Brown C; Canadian Thoracic Society COPD Committee Dyspnea Expert Working Group. Managing dyspnea in patients with advanced chronic obstructive pulmonary disease: a Canadian Thoracic Society clinical practice guideline. Can Respir J. 2011 Mar-Apr;18(2):69-78. doi: 10.1155/2011/745047. PMID 21499589
- [Background] 8. Global Initiative for Chronic Obstructive Lung Disease (GOLD). Global Strategy for the Diagnosis, Management and Prevention of COPD. 2022.
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Tsutsui M, Gerayeli F, Sin DD. Pulmonary Rehabilitation in a Post-COVID-19 World: Telerehabilitation as a New Standard in Patients with COPD. Int J Chron Obstruct Pulmon Dis. 2021 Feb 19;16:379-391. doi: 10.2147/COPD.S263031. eCollection 2021. PMID 33642858
- [Background] Cameron-Tucker HL, Wood-Baker R, Joseph L, Walters JA, Schuz N, Walters EH. A randomized controlled trial of telephone-mentoring with home-based walking preceding rehabilitation in COPD. Int J Chron Obstruct Pulmon Dis. 2016 Aug 25;11:1991-2000. doi: 10.2147/COPD.S109820. eCollection 2016. PMID 27601892
- [Background] Malaguti C, Dal Corso S, Janjua S, Holland AE. Supervised maintenance programmes following pulmonary rehabilitation compared to usual care for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2021 Aug 17;8(8):CD013569. doi: 10.1002/14651858.CD013569.pub2. PMID 34404111
- [Background] 13. World Health Organization. WHO-ITU Global Standard for Accessibility of Telehealth Services. . 2022.
- [Background] Ku BPS, Tse AWS, Pang BCH, Cheung NT, Pang JYW, Chan JKY, Hui HL, Chu D, Choi KHW. Tele-Rehabilitation to Combat Rehabilitation Service Disruption During COVID-19 in Hong Kong: Observational Study. JMIR Rehabil Assist Technol. 2021 Aug 19;8(3):e19946. doi: 10.2196/19946. PMID 34254945
- [Background] Zanaboni P, Dinesen B, Hjalmarsen A, Hoaas H, Holland AE, Oliveira CC, Wootton R. Long-term integrated telerehabilitation of COPD Patients: a multicentre randomised controlled trial (iTrain). BMC Pulm Med. 2016 Aug 22;16(1):126. doi: 10.1186/s12890-016-0288-z. PMID 27549782
- [Background] Zanaboni P, Lien LA, Hjalmarsen A, Wootton R. Long-term telerehabilitation of COPD patients in their homes: interim results from a pilot study in Northern Norway. J Telemed Telecare. 2013 Oct;19(7):425-9. doi: 10.1177/1357633X13506514. PMID 24218358
- [Background] Cerdan-de-Las-Heras J, Balbino F, Lokke A, Catalan-Matamoros D, Hilberg O, Bendstrup E. Effect of a New Tele-Rehabilitation Program versus Standard Rehabilitation in Patients with Chronic Obstructive Pulmonary Disease. J Clin Med. 2021 Dec 21;11(1):11. doi: 10.3390/jcm11010011. PMID 35011755
- [Background] Bernocchi P, Vitacca M, La Rovere MT, Volterrani M, Galli T, Baratti D, Paneroni M, Campolongo G, Sposato B, Scalvini S. Home-based telerehabilitation in older patients with chronic obstructive pulmonary disease and heart failure: a randomised controlled trial. Age Ageing. 2018 Jan 1;47(1):82-88. doi: 10.1093/ageing/afx146. PMID 28985325
- [Background] Crisafulli E, Clini EM. Measures of dyspnea in pulmonary rehabilitation. Multidiscip Respir Med. 2010 Jun 30;5(3):202-10. doi: 10.1186/2049-6958-5-3-202. PMID 22958431
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Background] Lapin BR, Kinzy TG, Thompson NR, Krishnaney A, Katzan IL. Accuracy of Linking VR-12 and PROMIS Global Health Scores in Clinical Practice. Value Health. 2018 Oct;21(10):1226-1233. doi: 10.1016/j.jval.2018.03.011. Epub 2018 Apr 26. PMID 30314624
- [Background] Schalet BD, Rothrock NE, Hays RD, Kazis LE, Cook KF, Rutsohn JP, Cella D. Linking Physical and Mental Health Summary Scores from the Veterans RAND 12-Item Health Survey (VR-12) to the PROMIS((R)) Global Health Scale. J Gen Intern Med. 2015 Oct;30(10):1524-30. doi: 10.1007/s11606-015-3453-9. Epub 2015 Jul 16. PMID 26179820
- [Background] Formiga MF, Roach KE, Vital I, Urdaneta G, Balestrini K, Calderon-Candelario RA, Campos MA, Cahalin LP. Reliability and validity of the test of incremental respiratory endurance measures of inspiratory muscle performance in COPD. Int J Chron Obstruct Pulmon Dis. 2018 May 15;13:1569-1576. doi: 10.2147/COPD.S160512. eCollection 2018. PMID 29805255
- [Background] COPD Foundation. COPD Foundation Educational Materials. In:2023.
- [Background] Ross RM, Murthy JN, Wollak ID, Jackson AS. The six minute walk test accurately estimates mean peak oxygen uptake. BMC Pulm Med. 2010 May 26;10:31. doi: 10.1186/1471-2466-10-31. PMID 20504351
- [Background] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406
- [Background] Beaumont M, Mialon P, Le Ber C, Le Mevel P, Peran L, Meurisse O, Morelot-Panzini C, Dion A, Couturaud F. Effects of inspiratory muscle training on dyspnoea in severe COPD patients during pulmonary rehabilitation: controlled randomised trial. Eur Respir J. 2018 Jan 25;51(1):1701107. doi: 10.1183/13993003.01107-2017. Print 2018 Jan. PMID 29371379
- [Background] de Souza E Silva CG, Kaminsky LA, Arena R, Christle JW, Araujo CGS, Lima RM, Ashley EA, Myers J. A reference equation for maximal aerobic power for treadmill and cycle ergometer exercise testing: Analysis from the FRIEND registry. Eur J Prev Cardiol. 2018 May;25(7):742-750. doi: 10.1177/2047487318763958. Epub 2018 Mar 8. PMID 29517365
- [Background] Billinger SA, VAN Swearingen E, McClain M, Lentz AA, Good MB. Recumbent stepper submaximal exercise test to predict peak oxygen uptake. Med Sci Sports Exerc. 2012 Aug;44(8):1539-44. doi: 10.1249/MSS.0b013e31824f5be4. PMID 22382170
- [Background] Herda AA, Lentz AA, Mattlage AE, Sisante JF, Billinger SA. Cross-validation of the recumbent stepper submaximal exercise test to predict peak oxygen uptake in older adults. Phys Ther. 2014 May;94(5):722-9. doi: 10.2522/ptj.20130307. Epub 2014 Jan 16. PMID 24435104
- [Derived] Karim R, Smith L, Baldwin J, Pham R, Kim HJ, Miccile L, Sullivan M, Gore S. Comparison of Telehealth and Onsite Supervised Maintenance Exercise Programs for Adults With Chronic Lung Disease: Protocol for a Pilot Randomized Feasibility Trial. JMIR Res Protoc. 2025 Aug 25;14:e71039. doi: 10.2196/71039. PMID 40854211